CLINICAL TRIAL: NCT02243592
Title: Exceptional Responders Pilot Study: Molecular Profiling of Tumors From Cancer Patients Who Are Exceptional Responders
Brief Title: Molecular Profiling in Tissue Samples From Patients With Cancer Who Are Exceptional Responders to Treatment
Status: Active, not recruiting | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: NCI-2014-01585; NCI-2014-01585 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9671 (Other: National Cancer Institute); 9671 (Other: CTEP); UM1CA186704 (NIH); NCT02496195 (obsolete NCT alias)
Record Dates: First submitted 2014-09-16; First posted 2014-09-18 (Estimated); Last update posted 2026-02-12 (Actual); Status verified 2025-09

CONDITIONS: Malignant Neoplasm
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Tissue, blood, and buccal cells
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Ancillary-Correlative (molecular profiling): Previously collected tissue samples are analyzed via whole exome sequencing and/or targeted NGS assay deep sequencing. Cases for which sufficient nucleic acid amounts are available will undergo additional analyses including whole genome sequencing, mRNA-sequencing, miRNA sequencing, promoter methylation analysis, and SNP analysis.
  Interventions: Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Undergo sequencing and SNP analysis

SUMMARY:
This pilot research trial studies molecular profiling in tissue samples from patients with cancer who got better with treatment that didn't work for most other patients with the same disease. Studying samples of tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in deoxyribonucleic acid (DNA) and identify biomarkers related to how well patients respond to treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To identify molecular indicators in malignant tissues from patients who were exceptional responders on clinical trials or standard systemic treatments using whole exome and/or targeted deep sequencing, as well as potentially other sequencing and other molecular characterization methods (if adequate tissue exists).

II. To explore associations between the identified molecular indicators and the putative mechanism of action of the treatment received by the patient.

III. To test the feasibility of identifying "exceptional responders", obtaining the relevant tumor and normal tissue and clinical data, and performing whole exome and/or targeted deep sequencing on these samples.

OUTLINE:

Previously collected tissue samples are analyzed via whole exome sequencing and/or targeted next generation sequencing (NGS) assay deep sequencing. Cases for which sufficient nucleic acid amounts are available will undergo additional analyses including whole genome sequencing, messenger ribonucleic acid (RNA) (mRNA)-sequencing, micro (miRNA) sequencing, promoter methylation analysis, and single nucleotide polymorphism (SNP) analysis.

ELIGIBILITY:
Inclusion Criteria:

* Documented exceptional response, defined as patients meeting the following criteria:

  * Complete response to a regimen in which complete response is expected in < 10% of similarly treated patients
  * Partial response (PR) > 6 months in a regimen in which PRs > 6 months are expected in < 10% of patients with similar disease treated with same or similar regimen
  * Complete response (CR) or PR of unusual duration, such that the internal review committee considers it to be an exceptional response; examples below:

    * PR of duration > 3 x the median expected PR duration (in cases where PR is expected in > 10% of patients with the same disease treated with the same regimen)
    * CR or duration > 3 x the median expected CR duration (in cases where CR may be seen in > 10% of patients with same disease treated with same regimen)
    * The observed duration of CR (or PR) is longer than expected for 90% of patients with same disease treated with same regimen
  * Note: it is not required that the patient be enrolled on a clinical trial when the exceptional response was observed
* Reports of radiologic scans or other evidence documenting response will be submitted for review; cases where response is not assessable (e.g. adjuvant treatment) will not be eligible because the outcome can not be attributed to a specific treatment
* Treatment history must be available, for prior treatment and for the drug to which the exceptional response occurred
* Patient must meet consent criteria; this requires: (i) current exceptional responder (ER) consent by a living participant not lost to follow-up, (ii) prior consent for future research by a participant not known to be deceased, but lost to follow-up, or (iii) if patient is deceased and did not decline to participate in research at the time of tissue removal for any tissue that would be used in this study, then no consent is required
* Tumor sample available that meets study requirements
* Required tumor samples MUST exist and be able to be submitted; investigators wishing to submit samples must not have made agreements that would prohibit the free use of data from such samples; the National Cancer Institute (NCI) will provide investigators with a letter for the collaborator amending their existing agreement to allow for the case to be submitted

  * Tumor tissue from prior to administration of the drug to which the exceptional response occurred is required; ideally this sample will have been collected just prior to treatment, but other prior tissue will be considered; tissue may be fresh frozen or formalin-fixed paraffin embedded
  * Tumor tissue amount must be at least a core biopsy, and meet minimum specimen requirements
* Encouraged: normal tissue sample: (optional): blood or other specimen source for germline sequencing
* The tumor samples and clinical data submitted to the Exceptional Responders Database in database in Genotypes and Phenotypes (dbGaP) will need to have appropriate agreements in place to allow for the submission; the Exceptional Responders Database can accept clinical data and samples from cases enrolled on a Cancer Therapy Evaluation Program (CTEP) sponsored clinical trial and cases that were not enrolled on any clinical trial; if the response occurred on a trial that was not CTEP-sponsored, there are existing agreements between the submitting site and the pharmaceutical company; if existing agreements do not allow for the submission of sample and clinical data, the NCI will provide the investigators with a letter that allows the tissue to be used for the exceptional responders study if signed by the appropriate collaborator; the letter modifies the existing agreement to include the CTEP Intellectual Property (IP) Option language that would allow the case to be submitted to the Exceptional Responders Database; if the existing agreement cannot be modified and the letter cannot be signed, the proposed case will not be accepted; Note: as stated above, the patient does not need to have been enrolled on a clinical trial to be eligible for the exceptional responders study

Exclusion Criteria:

* Patient's response did not meet criteria for an exceptional response
* Patient's treatment regimen is expected to lead to CR or durable PR in > 10% of patients
* Patient's duration of response is not > 3 x expected median length of response
* Response not evaluable or not able to be attributed to systemic treatment (e.g. adjuvant treatment)
* Patient refused consent for use of tissue for research activities included in the exceptional responders study
* Tumor sample from prior to the exceptional response is not available, or does not meet quality metrics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with cancer participating in the Exceptional Cases Initiative
Sampling Method: Non-Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2014-09-24 (Actual); Primary Completion 2021-03-04 (Actual); Study Completion 2026-04-02 (Estimated)

PRIMARY OUTCOMES:
Molecular features in tissue samples from patients who were exceptional responders | Baseline
  The molecular features of the tumors in the patients will be discernible as distinct to the tumor by comparison to (i) samples from normal tissue in the same patient and (ii) databases of similar data for normal and other tumor types.
Putative mechanisms of action of the treatments that the patients received when they experienced their exceptional responses | Baseline
  The associations between identified molecular features and the putative mechanisms of action of the treatments that the patients received when they experienced their exceptional responses will be explored. Statistical analyses will be primarily descriptive.
Number of cases identified as potential exceptional responders | Baseline
  Statistical analyses will be primarily descriptive.
Percentage of identified potential cases confirmed to be exceptional responders | Baseline
  Statistical analyses will be primarily descriptive.
Percentage of confirmed exceptional responders for which adequate tissue with appropriate informed consent is acquired | Baseline
  Statistical analyses will be primarily descriptive.
Percentage of acquired cases with tissue for which at least the minimum molecular characterization is successfully obtained | Baseline
  Statistical analyses will be primarily descriptive.
Percentage of molecularly characterized cases for which a Molecular Characterization report identified (without reference to the drug received by the patient) at least one feature judged to have potential therapeutic relevance | Baseline
  Promising discoveries will be summarized for the group of cases for which the minimum molecular characterization was successfully obtained. For each such case, molecular data will be reviewed by an expert panel ("Panel") to identify interesting features. All estimated proportions will be accompanied by exact 95% confidence intervals.
Percentage of cases with >= 1 feature on Molecular Characterization report that was judged to have potential therapeutic relevance to the specific class of drug the patient actually received when the exceptional response was experienced | Baseline
  Promising discoveries will be summarized for the group of cases for which the minimum molecular characterization was successfully obtained. For each such case, molecular data will be reviewed by the Panel to identify interesting features. All estimated proportions will be accompanied by exact 95% confidence intervals.
Percentage of cases with >= 1 feature that correlates with the mechanism of action of the specific grant to which the exceptional response occurred that was found after further analyzing the molecular profile data for relevant molecular abnormalities | Baseline
  Promising discoveries will be summarized for the group of cases for which the minimum molecular characterization was successfully obtained. For each such case, molecular data will be reviewed by the Panel to identify interesting features. All estimated proportions will be accompanied by exact 95% confidence intervals.

CONTACTS AND LOCATIONS:
Overall Officials: S. P Ivy, Principal Investigator — National Cancer Institute (NCI)
Locations (73):
- United States (73):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Kaiser Permanente-Fresno, Fresno, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Kaiser Permanente-Richmond, Richmond, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Greenwich Hospital, Greenwich, Connecticut
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - John B Amos Cancer Center, Columbus, Georgia
  - South Georgia Medical Center/Pearlman Cancer Center, Valdosta, Georgia
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Rush MD Anderson Cancer Center, Chicago, Illinois
  - Presence Resurrection Medical Center, Chicago, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Physicians' Clinic of Iowa PC, Cedar Rapids, Iowa
  - York Hospital, York Village, Maine
  - National Cancer Institute Developmental Therapeutics Clinic, Bethesda, Maryland
  - NCI - Center for Cancer Research, Bethesda, Maryland
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - UP Health System Hematology Oncology Marquette, Marquette, Michigan
  - UP Health System Marquette, Marquette, Michigan
  - Henry Ford Health Providence Southfield Hospital, Southfield, Michigan
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Portsmouth Regional Hospital, Portsmouth, New Hampshire
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - University of Rochester, Rochester, New York
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Riverside Methodist Hospital, Columbus, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Kaiser Permanente Northwest, Portland, Oregon
  - Reading Hospital McGlinn Cancer Institute at Phoenixville, Phoenixville, Pennsylvania
  - Chester County Hospital, West Chester, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Wellmont Holston Valley Hospital and Medical Center, Kingsport, Tennessee
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Ben Taub General Hospital, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - WVUH-Berkely Medical Center, Martinsburg, West Virginia
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin

REFERENCES:
- [Derived] Moore KN, Mannel RS. Is the NCI MATCH trial a match for gynecologic oncology? Gynecol Oncol. 2016 Jan;140(1):161-6. doi: 10.1016/j.ygyno.2015.11.003. Epub 2015 Nov 14. PMID 26586415